CLINICAL TRIAL: NCT04361032
Title: Assessment of Efficacy and Safety of Tocilizumab Compared to DefeROxamine, Associated With Standards Treatments in COVID-19 (+) Patients Hospitalized In Intensive Care in Tunisia. Multicentric, Comparative, Randomized Study
Brief Title: Assessment of Efficacy and Safety of Tocilizumab Compared to DefeROxamine, Associated With Standards Treatments in COVID-19 (+) Patients Hospitalized In Intensive Care in Tunisia
Acronym: TRONCHER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abderrahmane Mami Hospital (Other)
Collaborators: Eshmoun Clinical Research Center (Network); Datametrix (Industry)
Responsible Party: Principal Investigator, Dr Jalila Ben Khelil, Head of department, Abderrahmane Mami Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECC2020-06
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: COVID19; Intensive Care Unit
Keywords: Deferoxamine; Tocilizumab
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): ROACTEMRA: (8mg/ kg per day) (1 injection per infusion)
  Interventions: Drug: Tocilizumab Injection
- Deferoxamine (Active Comparator): DESFERAL: 500 mg, powder, and solvent for IV solution
  Interventions: Drug: Deferoxamine

INTERVENTIONS:
Drug: Tocilizumab Injection — Tocilizumab (LOC) (8mg/ kg per day) (1 injection per infusion). Only on the 1st day (D0)
  Other Names: ROACTEMRA
  Arms: Tocilizumab
Drug: Deferoxamine — Deferoxamine (Desferal 500 mg, powder, and solvent for IV solution for injection)
  Other Names: DESFERAL
  Arms: Deferoxamine

SUMMARY:
Assessment of Efficacy and Safety of Tocilizumab Compared to DefeROxamine, associated with standards treatments in COVID-19 (+) patients, Hospitalized In Intensive care in Tunisia.

Multicentric, comparative, randomized study.

DETAILED DESCRIPTION:
Arm1 :

* Usual standard treatment*
* Tocilizumab (LOC) (8mg/ kg per day) (1 injection per infusion) a second injection may be considered if necessary, but no more than 800 mg per day. Only on the 1st day (D0)
* Enoxaparin (4000 IU X 2) per day for the duration of hospitalization

VERSUS

Arm 2:

* Usual standard treatment*
* Deferoxamine (Desferal 500 mg, powder, and solvent for IV solution) by electric syringe 40 mg/kg/day 5day/7 without exceeding 5 g per day for 14 days
* Enoxaparin (4000 IU X 2) per day for the duration of hospitalization

Usual standard treatment*: according to the standard practices of each center, apart from the active molecules of the 2 arms and their therapeutic class)

ELIGIBILITY:
Inclusion Criteria:

* Patient confirmed COVID19 positive
* Patient with acute respiratory deficiency
* Patient hospitalized in the intensive care unit
* Age >18 years old
* Having given written consent for their participation in the study

Exclusion Criteria:

* Taking Tocilizumab or hydroxychloroquine deferoxamine within one month prior to inclusion (excluding participation in THINC or COVID_2Pro or COVID+PA studies)
* Severe/severe liver failure
* Dialysis patients
* Renal insufficiency (clearance< 30ml/min/1.73m2)
* Allergy to deferoxamine
* Pregnant or breastfeeding woman
* Hypersensitivity to the active substance or any of the excipients of Tocilizumab
* A decrease in blood platelets with previous use of enoxaparin or another heparin drug,
* hemophilia and related diseases,
* stomach or duodenal ulcer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-09-04 (Estimated); Primary Completion 2020-09-04 (Estimated); Study Completion 2020-10-04 (Estimated)

PRIMARY OUTCOMES:
the mortality rate | 90 day
  * Evaluate the mortality rate at 90 days.
  * Evaluate the Intensive Care Unit (ICU) and Hospital Mortality rate at day 90 with date and cause of death (if applicable)

CONTACTS AND LOCATIONS:
Locations (1):
- Eshmoun Clinical Research Centre/ Hôpital Abderrahmane Mami-Ariana, Aryanah, Tunisia

IPD SHARING:
Plan to Share IPD: No